CLINICAL TRIAL: NCT01728727
Title: Safety and Efficacy of Human Umbilical Cord Derived Mesenchymal Stem Cells for Treatment of HBV-related Liver Cirrhosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other); Eastern Hepatobiliary Surgery Hospital (Other); Chinese Academy of Medical Sciences (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Han Ying, professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120912-3
Record Dates: First submitted 2012-10-31; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Liver Cirrhosis; End Stage Liver Disease
Keywords: liver cirrhosis; end stage liver disease; umbilical cord; mesenchymal stem cells; HBV
MeSH Terms: conditions — Liver Cirrhosis; End Stage Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional (Active Comparator): conventional treatment & antiviral treatment
  Interventions: Other: conventional treatment
- UC-MSC transplantation (Experimental): Participants will receive umbilical cord derived mesenchymal stem cell treatment at day 1 and conventional treatment and antiviral treatment through the one year study visit. Participants will then be followed until one years study visit
  Interventions: Other: UC-MSC transplantation

INTERVENTIONS:
Other: UC-MSC transplantation — After enrolled, Participant will receive umbilical cord MSC transplantation of 1*10E6 cells/kg via hepatic artery. Participant will then be followed until 1 years study visit
  Arms: UC-MSC transplantation
Other: conventional treatment — Participants will receive conventional treatment and antiviral treatment.
  Arms: conventional

SUMMARY:
HBV related Liver disease is a common medical problem in China. An estimated 7.18% of the Chinese (about 93 million) is infected with hepatitis B, and most of the HBV- related hepatitis can developed into liver cirrhosis.

Liver transplantation is the only available life saving treatment for patients with end stage liver disease. However, lack of donors, surgical complications, rejection, and high cost are serious problems.

Mesenchymal stem cells (MSCs) possess plasticity and have the potential to differentiate into hepatocyte; Thus, MSCs hold great hope for therapeutic applications. Human umbilical cord-derived MSCs (hUC-MSCs) exhibit a more beneficial immunogenic profile and greater overall immunosuppressive potential than aged bone marrow-derived MSCs. Like MSCs derived from bone marrow, hUC-MSCs can also be used to treat rat liver fibrosis and improve glucose homeostasis in rats with liver cirrhosis. In this study, the patients with HBV-related liver cirrhosis will undergo administration of hUC-MSCs via hepatic artery to evaluate the safety and efficacy of hUC-MSC treatment for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. HBV-related liver cirrhosis
3. Child-Pugh score 9-15
4. Written consent -

Exclusion Criteria:

1. Hepatocellular carcinoma or other malignancies
2. Severe problems in other vital organs(e.g.the heart,renal or lungs)
3. Pregnant or lactating women
4. Severe bacteria infection
5. Anticipated with difficulty of follow-up observation
6. Other candidates who are judged to be not applicable to this study by doctors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
one year survival rate | one year after treatment

SECONDARY OUTCOMES:
MELD score | 1week, 4weeks,3months, 6months, 9months and 1year after treatment
Child Pugh Score | 1week, 4weeks,3months, 6months, 9months and 1year after treatment
alpha fetoprotein | 1week, 4weeks,3months, 6months, 9months and 1year after treatment
renal function | 1week, 4weeks,3months, 6months, 9months and 1year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daiming Fan, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital of Digestive Disease, Xi'an, Shaanxi, China